CLINICAL TRIAL: NCT00317122
Title: Demonstrate Non-inferiority of GSK Biologicals' Tritanrix™-HepB/Hib-MenAC vs Tritanrix™-HepB/Hiberix™ With Respect to Anti-HBs Immune Response, When Given to Healthy Infants at 6,10 & 14 Weeks Age, After a Birth Dose of Hepatitis B Vaccine
Brief Title: Assess the Immune Response Following Primary Vaccination With GSK Biologicals' Tritanrix™-HepB/Hib-MenAC vs Tritanrix™-HepB/Hiberix™ Given at 6,10 & 14 Wks of Age to Infants Who Received Hepatitis B Vaccine at Birth
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 759346/007
Record Dates: First submitted 2006-02-23; First posted 2006-04-24 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Diphtheria; Haemophilus Influenzae Type b; Hepatitis B; Tetanus; Whole Cell Pertussis
MeSH Terms: conditions — Diphtheria; Haemophilus Infections; Hepatitis B; Tetanus

INTERVENTIONS:
Biological: DTPw-HBV/Hib-MenAC conjugate vaccine

SUMMARY:
This study will only include infants born to mothers who are tested as seronegative for human immunodeficiency virus (HIV) & hepatitis B surface antigen (HBsAg). The purpose of this study is to demonstrate in infants who received a birth dose of hepatitis B vaccine that Tritanrix™-HepB/Hib-MenAC vaccine is at least as good as Tritanrix™-HepB/Hiberix™ with respect to immunogenicity of the hepatitis B antigen.

DETAILED DESCRIPTION:
Randomized study with two groups to receive one of the following vaccination regimens:

* GSK Biologicals' Tritanrix™-HepB/Hib-MenAC
* GSK Biologicals' Tritanrix™-HepB/Hiberix™

ELIGIBILITY:
Inclusion criteria:

* Healthy infants aged 7 days +/- 3 days old born to mothers who are tested as seronegative for HIV & HBsAg, written informed consent obtained from the parents, born after a gestation period of 36 to 42 weeks.

Exclusion criteria:

* Known exposure to diphtheria, tetanus, pertussis, hepatitis B, Haemophilus influenzae type b and/or meningococcal disease since birth.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on physical examination.
* A family history of congenital or hereditary immunodeficiency.
* Major congenital defects or serious illness.
* Any neurologic disorders or seizures.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
* A birth dose of hepatitis B vaccine given outside the frame of this study.

Ages: 4 Days to 10 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 192 (Actual)
Dates: Start 2004-10; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
One month after the third dose of the primary vaccination, measurement of anti-HBs antibody concentrations.

SECONDARY OUTCOMES:
Immunogenicity: One month after the third dose of the primary vaccination, antibody concentrations or titres against all other vaccine antigens.
Reactogenicity and safety: after each dose: solicited (day 0-3, local & general) & unsolicited (day 0-30) symptoms. Over the full course of the study: serious adverse events (SAEs)"

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- South Africa (3):
  - GSK Investigational Site, Brits
  - GSK Investigational Site, Centurion
  - GSK Investigational Site, Ga-Rankuwa

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 759346/007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 759346/007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 759346/007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 759346/007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 759346/007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 759346/007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register